CLINICAL TRIAL: NCT00006760
Title: A Pilot Study of Re-Induction Chemotherapy With Ifosfamide, and Vinorelbine (IV) in Children With Refractory/Relapsed Hodgkin's Disease
Brief Title: Combination Chemotherapy in Treating Children With Refractory or Relapsed Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AHOD00P1; CCG-A5981 (Other: Children's Cancer Group); CDR0000068325 (Other: Clinical Trials.gov); NCI-2012-02366 (Other: NCI); U10CA098543 (NIH)
Record Dates: First submitted 2000-12-06; First posted 2003-01-27 (Estimated); Last update posted 2013-07-26 (Estimated); Status verified 2013-07

CONDITIONS: Lymphoma
Keywords: recurrent/refractory childhood Hodgkin lymphoma; childhood lymphocyte predominant Hodgkin lymphoma; childhood lymphocyte depletion Hodgkin lymphoma; childhood nodular sclerosis Hodgkin lymphoma; childhood mixed cellularity Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Recurrence; Hodgkin Disease | interventions — Filgrastim; Ifosfamide; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (ifosfamide, vinorelbine, filgrastim) (Experimental): Patients receive ifosfamide IV over 24 hours on days 1-4 and vinorelbine tartrate IV over 6-10 minutes on days 1 and 5. Patients also receive filgrastim (G-CSF) subcutaneously or IV over 15-30 minutes beginning 24-36 hours after completion of vinorelbine and continuing daily until blood counts recover. Treatment repeats at least every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity. Patients may receive a third course of therapy at the discretion of the investigator. Heavily pretreated, high-risk patients who achieve a complete response are eligible for stem cell transplantation. Patients undergo peripheral blood stem cell (PBSC) collection during hematopoietic recovery after the second course of chemotherapy. Patients with sufficient PBSCs collected may undergo PBSC transplantation on protocol COG-AHOD0121.
  Interventions: Biological: filgrastim; Drug: ifosfamide; Drug: vinorelbine tartrate

INTERVENTIONS:
Biological: filgrastim — subcutaneously or IV over 15-30 minutes beginning 24-36 hours after completion of vinorelbine and continuing daily until blood counts recover.
Drug: ifosfamide — V over 24 hours on days 1-4
Drug: vinorelbine tartrate — IV over 6-10 minutes on days 1 and 5.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as ifosfamide and vinorelbine, work in different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy in treating children who have refractory or relapsed Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate (overall and within strata) in both minimally pretreated, low-risk and heavily pretreated, high-risk children with refractory or relapsed Hodgkin's lymphoma treated with ifosfamide and vinorelbine with filgrastim (G-CSF).
* Determine the cardiac, hepatic, renal, and hematologic toxicity of this regimen in minimally-pretreated, low-risk patients.
* Determine the toxic death rate in minimally pretreated, low-risk patients treated with this regimen.
* Determine whether this treatment regimen can mobilize sufficient hematopoietic stem cells (CD34) for subsequent stem cell transplantation in minimally pretreated, low-risk patients.
* Determine the incidence of hypermutability by longitudinal genotoxic biomonitoring of patients treated with this regimen.
* Determine the prognostic significance of biological markers, including serum interleukin (IL)-10 receptor, serum IL-2 receptor, p53, and mdm-2 in patients treated with this regimen.

OUTLINE: This is a multicenter study. Patients are stratified by prior therapy (minimally pretreated, low-risk vs heavily pretreated, high-risk).

Patients receive ifosfamide IV over 24 hours on days 1-4 and vinorelbine IV over 6-10 minutes on days 1 and 5. Patients also receive filgrastim (G-CSF) subcutaneously or IV over 15-30 minutes beginning 24-36 hours after completion of vinorelbine and continuing daily until blood counts recover. Treatment repeats at least every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity. Patients may receive a third course of therapy at the discretion of the investigator.

Heavily pretreated, high-risk patients who achieve a complete response are eligible for stem cell transplantation. Patients undergo peripheral blood stem cell (PBSC) collection during hematopoietic recovery after the second course of chemotherapy. Patients with sufficient PBSCs collected may undergo PBSC transplantation on protocol COG-AHOD0121.

Patients are followed at 1, 6, and 12 months and then periodically thereafter.

PROJECTED ACCRUAL: A total of 66 patients will be accrued for this study within 1.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed refractory or relapsed Hodgkin's lymphoma

  * Mixed cellularity, not otherwise specified (NOS)
  * Lymphocytic depletion, NOS
  * Lymphocytic depletion, diffuse fibrosis
  * Lymphocytic depletion, reticular
  * Lymphocytic predominance, NOS
  * Lymphocytic predominance, diffuse
  * Lymphocytic predominance, nodular
  * Hodgkin's paragranuloma NOS
  * Hodgkin's granuloma
  * Hodgkin's sarcoma
  * Nodular sclerosis, NOS
  * Nodular sclerosis, cellular phase
  * Nodular sclerosis, lymphocytic predominance
  * Nodular sclerosis, mixed cellularity
  * Nodular sclerosis, lymphocytic depletion
  * Other (type not specified)
* In first relapse
* Metastasis to bone marrow with granulocytopenia, anemia, and/or thrombocytopenia allowed
* Not enrolled on POG-9426 unless there is an extranodal site of recurrence

PATIENT CHARACTERISTICS:

Age:

* Under 30 at diagnosis

Performance status:

* Lansky 60-100% (for patients 16 years and under)
* Karnofsky 60-100% (for patients over 16 years)

Life expectancy:

* At least 2 months

Hematopoietic:

* See Disease Characteristics
* Absolute neutrophil count at least 1,000/mm^3
* Platelet count at least 75,000/mm^3 (transfusion independent)

Hepatic:

* Bilirubin no greater than 1.5 times normal
* SGOT or SGPT less than 2.5 times normal

Renal:

* Creatinine no greater than 1.5 times normal
* Creatinine clearance or radioisotope glomerular filtration rate at least 70 mL/min

Cardiovascular:

* Shortening fraction at least 27% by echocardiogram OR
* Ejection fraction at least 50% by gated radionuclide

Other:

* No other concurrent serious illness
* No known hypersensitivity to E. coli-derived proteins, filgrastim (G-CSF), or any other component of study drugs

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent immunomodulating agents

Chemotherapy:

* At least 2 weeks since prior chemotherapy (3 weeks for nitrosoureas) and recovered
* No other concurrent anticancer chemotherapy

Endocrine therapy:

* No concurrent steroids
* No concurrent corticosteroids (e.g., dexamethasone)

Radiotherapy:

* Recovered from prior radiotherapy

Surgery:

* Not specified

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 66 (Actual)
Dates: Start 2001-05; Primary Completion 2005-07 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Overall response rate | After 2 cycles
  Overall response includes complete response (CR) or partial response (PR).

SECONDARY OUTCOMES:
Rate of successful PBSC harvest during re-induction defined as the ability to harvest 5 x 10^6 CD34+ cells/kg | After 2 cycles
  Will be calculated.
Biologic markers | At enrollment and during/after therapy
Cardiac, hepatic, renal, hematologic toxicity | Within 1 month of completion of therapy
Toxic death | Within 1 month of Completion of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Trippett, MD, Study Chair — Memorial Sloan Kettering Cancer Center; Pedro A. de Alarcon, MD, Study Chair — St. Jude Children's Research Hospital
Locations (114):
- United States (101):
  - Comprehensive Cancer Center at University of Alabama at Birmingham, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Southern California Permanente Medical Group, Downey, California
  - Jonathan Jaques Children's Cancer Center at Miller Children's Hospital, Long Beach, California
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - Children's Hospital Central California, Madera, California
  - Children's Hospital of Orange County, Orange, California
  - Sutter Cancer Center, Sacramento, California
  - Kaiser Permanente Medical Center - Oakland, Sacramento, California
  - Children's Hospital and Health Center - San Diego, San Diego, California
  - Stanford Cancer Center at Stanford University Medical Center, Stanford, California
  - Children's Hospital Cancer Center, Denver, Colorado
  - Carole and Ray Neag Comprehensive Cancer Center at the University of Connecticut Health Center, Farmington, Connecticut
  - Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lee Cancer Care of Lee Memorial Health System, Fort Myers, Florida
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - Miami Children's Hospital, Miami, Florida
  - Florida Hospital Cancer Institute at Florida Hospital Orlando, Orlando, Florida
  - M.D. Anderson Cancer Center - Orlando, Orlando, Florida
  - Sacred Heart Cancer Center at Sacred Heart Hospital, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - St. Joseph's Cancer Institute at St. Joseph's Hospital, Tampa, Florida
  - Kaplan Cancer Center at St. Mary's Medical Center, West Palm Beach, Florida
  - Curtis & Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - St. Luke's Mountain States Tumor Institute - Boise, Boise, Idaho
  - University of Illinois Cancer Center, Chicago, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - St. Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Kosair Children's Hospital, Louisville, Kentucky
  - Children's Hospital of New Orleans, New Orleans, Louisiana
  - CancerCare of Maine at Eastern Maine Medial Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - Alvin and Lois Lapidus Cancer Institute at Sinai Hospital, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Spectrum Health Cancer Care - Butterworth Campus, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - Children's Hospital of Minnesota - Minneapolis, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Keesler Medical Center - Keesler Air Force Base, Keesler Air Force Base, Mississippi
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - Children's Mercy Hospital, Kansas City, Missouri
  - Hackensack University Medical Center Cancer Center, Hackensack, New Jersey
  - St. Barnabas Medical Center, Livingston, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Brooklyn Hospital Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Cancer Institute at New York University Medical Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Long Island Cancer Center at Stony Brook University Hospital, Stony Brook, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Children's Medical Center - Dayton, Dayton, Ohio
  - Toledo Hospital, Toledo, Ohio
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Institute of Oncology at Vilnius University, Portland, Oregon
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Greenville Hospital System Cancer Center, Greenville, South Carolina
  - T.C. Thompson Children's Hospital, Chattanooga, Tennessee
  - Texas Tech University Health Sciences Center School of Medicine, Amarillo, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - Baylor University Medical Center - Houston, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - INOVA Fairfax Hospital, Fairfax, Virginia
  - Children's Hospital of the King's Daughters, Norfolk, Virginia
  - Massey Cancer Center at Virginia Commonwealth University, Richmond, Virginia
  - Carilion Cancer Center of Western Virginia, Roanoke, Virginia
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - Madigan Army Medical Center - Tacoma, Tacoma, Washington
  - Edwards Comprehensive Cancer Center at Cabell Huntington Hospital, Huntington, West Virginia
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Australia (3):
  - Prince of Wales Private Hospital, Randwick, New South Wales
  - Westmead Institute for Cancer Research at Westmead Hospital, Westmead, New South Wales
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (10):
  - Alberta Children's Hospital, Calgary, Alberta
  - Children's & Women's Hospital of British Columbia, Vancouver, British Columbia
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Montreal Children's Hospital at McGill University Health Center, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Ste-Foy, Quebec
  - Allan Blair Cancer Centre at Pasqua Hospital, Regina, Saskatchewan
  - Saskatoon Cancer Centre at the University of Saskatchewan, Saskatoon, Saskatchewan